CLINICAL TRIAL: NCT04015466
Title: Advanced GC Multi-omic Characterization in EU and CELAC Populations
Acronym: LEGACY-2
Status: Completed | Type: Observational
Sponsor: Fundación para la Investigación del Hospital Clínico de Valencia (Other)
Collaborators: Instituto Nacional de Cancerologia de Mexico (Other); Amsterdam UMC, location VUmc (Other); Pontificia Universidad Catolica de Chile (Other); Vall d'Hebron Institute of Oncology (Other); INSTITUTO ALEXANDER FLEMING (Unknown); Hospital Central del IPS (Other); IPATIMUP - Instituto De Patologia E Imunologia Molecular Da Universidade Do Porto (Other)
Responsible Party: Sponsor
Other Study IDs: LEGACY-2
Record Dates: First submitted 2019-06-05; First posted 2019-07-11 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Gastric Cancer
Keywords: Gastric Cancer; Personalized medicine; Oncology; Solid tumor; Primary Intervention
MeSH Terms: conditions — Stomach Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumour Blood Stool Urine Nail
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Patients with high diagnostic suspicion of advanced GC diagnosis
- Control: Patients with confirmed absent of GC

SUMMARY:
Observational study (cohort type) of advanced GC patients that will be recruited prospectively to study biological factors associated with the disease and relevant clinical outcomes.

DETAILED DESCRIPTION:
Despite of multiple attempts to improve treatment in recent decades, none strategies has improved prognosis in locally advanced stage III and IV GC. A therapeutic approach to GC based on current histological and image criteria (Tumour Node Metastasis -TNM- stage) is insufficient. Although multiple targeted agents are currently under investigation, so far, only trastuzumab and ramucirumab have demonstrated efficacy in advanced GC and have a regulatory approval. For this reason, the identification of specific targets that could be susceptible for drug inhibition, is an urgent requirement. Moreover, most studies and current international databases on late-stage/advanced GC are largely based on Asian populations, in sharp contrast tumour biology and genome of EU or CELAC populations remain poorly known.

The primary objective of this study are to:

1. Characterize a multi-centric cohort including EU and CELAC populations diagnosed with advanced GC through a multi-omic approach including proteomics, genomics, transcriptomics, microbiome and exposome analysis due to study the determinants of GC.
2. Identify the regional differences in EU and CELAC populations recruiting patients for this study for each omic characterization due to identify the high-risk group populations.
3. Identify and select from the multi-omic approach those biomarkers useful for the development of an algorithm to guide the therapeutic approach for advanced GC.

ELIGIBILITY:
Cases:

* Inclusion criteria:

  * Subjects ≥18 years old.
  * GC diagnosis stages III and IV (including gastroesophageal junction cancer) and/or a gastroscopy indication due to the high diagnostic suspicion of GC as part of the study of his disease.
  * Has given and signed the IC to participate in this study.
* Exclusion criteria:

  • Patients diagnosed with GC early disease (stage I and II) suitable for resectable strategy.
* Withdrawal criteria:

  * Patients initially recruited with high suspicion of GC diagnosis but not confirmed by the pathological report.

Controls:

* Inclusion criteria (only for microbiome analysis):

  * Subjects ≥18 years old.
  * Subjects to whom a gastroscopy is indicated within clinical care and is confirmed absent of GC in the same centres will be matched in age (+/- 10 years), gender and pertaining from the same region of the GC case.
  * Has given and signed the IC to participate in this study.
* Exclusion criteria:

  * Subjects from a different geographic area from the cases.
  * Patients with high suspicion of GC.
  * Patients with previous histopathologic diagnosis of peptic (gastric or duodenal) ulcer disease and/or atrophy or intestinal metaplasia.
  * Patients that have received antimicrobials during the 4 weeks period prior to the endoscopy.
  * Patients that have received proton pump inhibitors or H2-receptor antagonists, at least 2 weeks prior to the endoscopy

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: * Subjects >18 years old, with high diagnostic suspicion of advanced GC diagnosis (Stage III and IV)
  * Subjects >18 years old to whom a gastroscopy was indicated and confirmed absent of GC.
Sampling Method: Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2019-06-12 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Development of a new diagnostic algorithm for gastric cancer that includes molecular landscape, patient history, histopathological and environmental factors, personal microbiome and immune landscape | 3 years
  The project will look for an integrative diagnostic algorithm that incorporates multi-parameter inputs and apply artificial intelligence to provide more personalized risk estimates and which will form the basis for future development of a clinical tool

SECONDARY OUTCOMES:
Proteomic analysis of gastric cancer tissue | 3 years
  Determine the expression of certain proteins using ICH and ISH
Genomics (tumour next-generation sequencing) | 3 years
  Determine differences in the genetic mutational profile of different populations
Transcriptomics (Nanostring immune gene expression panel) | 3 years
  Determine differences in the genetic expression profile of different populations
Microbiota sequencing (including level of Epstein-Barr virus [EBV] DNA) | 3 years
  Determine differences in the microbiota profile of different populations
Dietary habits as assessed by a new study-specific questionnaire | 3 years
  Determine differences in dietary habits of different populations and its correlation with risk to develop gastric cancer
Biological risk factors as assessed through medical chart review | 3 years
  Determine differences in biological risk factors of different populations and its correlation with risk to develop gastric cancer
Daily routines as assessed by a new study-specific questionnaire | 3 years
  Determine differences daily routines of different populations and its correlation with risk to develop gastric cancer

CONTACTS AND LOCATIONS:
Locations (8):
- Instituto Alexander Fleming, Buenos Aires, Argentina
- Pontificia Universidad Católica de Chile, Santiago, Chile
- Instituto Nacional de Cancerología de México, México, Mexico
- VU Medical Centre, Amsterdam, Netherlands
- GenPat, Asunción, Paraguay
- Institute of Pathology and Immunology of University of Porto, Porto, Portugal
- Spain (2):
  - Vall d'Hebron Institut d'Oncologia, Barcelona
  - Hospital Clínico Univeristario de Valencia, Valencia

REFERENCES:
- [Derived] van Schooten TS, Derks S, Jimenez-Marti E, Carneiro F, Figueiredo C, Ruiz E, Alsina M, Molero C, Garrido M, Riquelme A, Caballero C, Lezcano E, O'Connor JM, Esteso F, Farres J, Mas JM, Lordick F, Vogt J, Cardone A, Girvalaki C, Cervantes A, Fleitas T; members of LEGACy consortium. The LEGACy study: a European and Latin American consortium to identify risk factors and molecular phenotypes in gastric cancer to improve prevention strategies and personalized clinical decision making globally. BMC Cancer. 2022 Jun 13;22(1):646. doi: 10.1186/s12885-022-09689-9. PMID 35692051